CLINICAL TRIAL: NCT00989495
Title: Single-blind Comprehensive Cohort Study Incorporating a Randomized Controlled Design on Bracing in AIS: A Feasibility Study
Brief Title: Comprehensive Cohort Study of Bracing for Adolescent Idiopathic Scoliosis (AIS): A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Scoliosis Research Society (Other)
Responsible Party: Principal Investigator, Dr Daniel Yee Tak FONG, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: dytfong; HKCTR-819 (Registry Identifier: Hong Kong Clinical Trials Registry)
Record Dates: First submitted 2009-10-01; First posted 2009-10-05 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: AIS
MeSH Terms: interventions — Braces

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Brace - Randomized (Experimental): Participants were randomized to be braced
  Interventions: Device: Brace
- Observation - Randomized (No Intervention): Participants were randomized to be observed only
- Brace - preference based (Experimental): Participants chose to be braced
  Interventions: Device: Brace
- Observation - preference-based (No Intervention): Participants chose to be observed only

INTERVENTIONS:
Device: Brace — Wearing a Thoraco-Lumbo-Sacral-Orthosis (TLSO) for a minimum of 20 hours per day
  Arms: Brace - Randomized; Brace - preference based

SUMMARY:
The purpose of this study is to gain initial experience and information for proper planning and conduct of a confirmatory study (a multi-centre single-blind comprehensive cohort study of bracing).

DETAILED DESCRIPTION:
The study has been completed.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of AIS
2. Age ≥10 years
3. Risser sign 0-2
4. Cobb's angle 20 deg to <25 deg with documented deterioration of at least 5 deg within the past 4 months (with a maximum of 10 days deviation), or 25 deg to <30 deg

Exclusion Criteria:

1. History of treatment of AIS
2. >= 1 year postmenarchal (for girls only)
3. Physical or mental disability to adhere to bracing
4. Diagnosis of musculoskeletal or development illness that might be responsible for the spinal curvature
5. Structural thoracic scoliosis with apex above T7 (Note these patients are not suitable for under-arm brace)
6. Difficulty to read, understand, and complete the study questionnaires
7. Any criteria, which, in the opinion of the investigator, suggests that the subject would not be compliant with the study protocol

Min Age: 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2008-10; Primary Completion 2011-03 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Time to >= 6 degree curve progression from baseline, Time to curve exceeding 45 degree, Time to surgery recommended/undertaken. | Baseline and every four months

SECONDARY OUTCOMES:
SRS-22 questionnaire, C-STAI questionnaire, C-BDI-II. | Baseline and every four months

CONTACTS AND LOCATIONS:
Overall Officials: Daniel YT Fong, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The Duchess of Kent Children's Hospital, Hong Kong, China